CLINICAL TRIAL: NCT06183762
Title: Real-World Treatment Patterns and Effectiveness of Targeted and Systemic Therapy in Patients With Advanced Lung Cancer Carrying MET Mutation-Positive
Brief Title: A Real-World Study of Treatment Patterns and Effectiveness in MET Mutation-Positive Advanced Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Other Study IDs: MET RWS
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ICIs: Patients receiving in first-line immunotherapy with or without anti-angiogenic or chemotherapy
  Interventions: Other: No treatment is included in this protocol.
- Savolitinib: Patients receiving in first-line savolitinib treatment
  Interventions: Other: No treatment is included in this protocol.
- Glumetinib: Patients receiving in first-line glumetinib treatment
  Interventions: Other: No treatment is included in this protocol.
- Bozitinib: Patients receiving in first-line bozitinib treatment
  Interventions: Other: No treatment is included in this protocol.

INTERVENTIONS:
Other: No treatment is included in this protocol. — No drug intervention or tissue sampling will be included in this study.

SUMMARY:
This is a descriptive observational study in which data are collected in an epidemiological manner. This study is not intended to alter or interfere with the current medical practice of the enrolled patients. Data will be collected in a forward-looking manner. This is a descriptive observational study in which data are collected in an epidemiological manner. This study is not intended to alter or interfere with the current medical practice of the enrolled patients. Data from patients on prior treatment will be collected retrospectively, and data from patients who will be treated later and included in the study will be collected in a prospective manner. The criteria for retrospective collection were consistent with those for prospective collection. Eligible patients will be enrolled after NGS analysis of tumor tissue and informed consent has been obtained. Information required for the study will be collected (every 3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 years of age.
2. Provision of fully informed consent prior to any study specific procedures.
3. Histologically or cytologically confirmed, unresectable stage IIIB/IIIC or stage IV NSCLC.
4. Genetic variants of tumor tissue detected by NGS.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced lung cancer, MET gene mutations
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | Assessed up to around 4.5 years
  From the time the first patient included in the observational analysis received treatment until disease progression, death due to various causes or censored at the date of last contact
Overall Survival | Assessed up to around 4.5 years
  From the time the first patient included in the observational analysis received treatment until death due to various causes or censored at the date of last contact

SECONDARY OUTCOMES:
Clinical relevance between genomic profiling and progression-free-survival | Assessed up to around 4.5 years
  Kaplan-Meier analysis for progression-free survival, utilizing data from various genetic testing methods including NGS and FISH, to evaluate the impact of different genetic alterations.
Clinical relevance between genomic profiling and overall survival | Assessed up to around 4.5 years
  Kaplan-Meier analysis for overall survival, utilizing data from various genetic testing methods including NGS and FISH, to evaluate the impact of different genetic alterations.
ORR | Assessed up to around 4.5 years
  Proportion of patients whose tumor volume shrinks to a pre-specified value (usually 30%) and who are able to maintain the minimum timeframe requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Province Tumor Hospital, Changsha, Hunan, China